CLINICAL TRIAL: NCT03101839
Title: A Phase I, Open-Label, Multicentre Dose-Escalation Study to Investigate the Safety and Pharmacokinetics of AZD4785 in Patients With Advanced Solid Tumours Where KRAS May Be an Important Driver of Tumour Survival
Brief Title: Phase I Dose-Escalation Study of AZD4785 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8360C00001; REFMAL 484 (Other: Sarah Cannon Development Innovations)
Record Dates: First submitted 2017-03-22; First posted 2017-04-05 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer; Advanced Solid Tumours
Keywords: AZD4785; KRAS; KRAS mutations; Non-small cell lung cancer; Advanced solid tumours
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD4785 (Experimental): This is a single-arm study in which all patients will receive AZD4785 by IV infusion. Patients will continue to receive treatment with AZD4785 until disease progression, intolerable toxicity, or discontinuation criteria are met.
  Interventions: Drug: AZD4785

INTERVENTIONS:
Drug: AZD4785 — KRAS Antisense Oligonucleotide

SUMMARY:
A Phase I, open-label, multicentre, dose-escalation study to investigate the safety, pharmacokinetics and maximum tolerated dose (MTD) of AZD4785 in patients with advanced solid tumours where KRAS may be an important driver of tumour survival.

Part A: Dose escalation in patients with solid tumours to evaluate safety, pharmacokinetics and maximum tolerated dose (MTD). Once the maximum tolerated dose (MTD) is established, a dose expansion cohort may be included in Part A, with up to an additional 6 patients to further explore the PK, safety, tolerability, and preliminary anti-tumour activity of the AZD4785 MTD for confirmation of the recommended phase 2 dose (RP2D).

Part B: Expansion cohort at the selected dose in patients with non-small cell lung cancer (NSCLC) to evaluate PK parameters, safety, tolerability, and preliminary anti-tumour activity of the AZD4785 RP2D as monotherapy in patients with NSCLC. Approximately 20 patients with NSCLC (Two groups of approximately 10 patients each) with NSCLC will be enrolled to Part B. Group 1 patients will have an option to provide tumour biopsies and Group 2 will be required (mandatory) to provide paired tumour biopsies. Overall up to 12 patients in Group 2Part B patients will be required (mandatory) to may provide paired tumour biopsies. A third group of up to 20 patients with other tumour types and/or a potential different schedule may be added based on the results seen in Parts A and B and any other emerging data and may also provide biopsies.

DETAILED DESCRIPTION:
This is a First-Time-in-Human (FTIH), Phase 1 study to determine the MTD, recommended Phase 2 dose (RP2D), safety, tolerability, pharmacodynamics, and pharmacokinetics of AZD4785. The study will be conducted in two parts: a dose-escalation phase (Part A)and an expansion phase (Part B). A third group of up to 20 patients with other tumour types and/or a potential different schedule may be added based on the results seen in Parts A and B and any other emerging data.

AZD4785 will be given as an IV infusion over 1 hour, initially in 3 loading doses during the first week and then weekly thereafter. The loading doses will be given on Days 1, 3, and 5 of the first week and weekly thereafter on Days 8, 15, and 22 of 28 Day cycles. In subsequent cycles AZD4785 will be administered on Days 1, 8, 15, and 22 until disease progression, intolerable toxicity, or discontinuation criteria have been met.

Once the MTD is established, a dose expansion cohort may be included in Part A, with up to 6 additional patients to explore the PK, safety, tolerability, and preliminary anti-tumour activity of the AZD4785 MTD for confirmation of the RP2D. Thereafter, Part B expansion phase will continue to explore PK parameters, safety, tolerability, and preliminary anti-tumour activity of the AZD4785 RP2D as monotherapy in patients with NSCLC. Approximately 20 patients with NSCLC (2 groups of approximately 10 patients each) with NSCLC will be enrolled to Part B. Group 1 patients will have an option to provide tumour biopsies and Group 2 will be required (mandatory) to provide paired tumour biopsies. Overall up to 12 patients in Part B may provide paired tumour biopsies. A third group of up to 20 patients with other tumour types and/or a potential different schedule may be added based on the results seen in Parts A and B and any other emerging data and may also provide biopsies. Up to 12 patients in Part B may provide paired biopsies.

ELIGIBILITY:
Inclusion Criteria

Part A Dose Escalation: Patients must have histological or cytological confirmation of a solid tumour known to harbour KRAS mutations (e.g., NSCLC, mCRC, pancreatic or cholangiocarcinoma), and have progressed despite standard therapy(ies), or are intolerant to standard therapy(ies), or have a tumour for which no standard therapy(ies) exists.

Part B Expansion: Patients in Part B must have measurable disease as measured by Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1

Group 1. Patients must have histological or cytological confirmation of locally advanced or metastatic KRASm+ NSCLC, who have failed prior therapy and for whom no current therapy is available.

Group 2. Patients must have histological or cytological confirmation of locally advanced or metastatic KRASm+ NSCLC, who have failed prior therapy and for whom no current therapy is available. At study entry patients must be clinically suitable for mandatory baseline and on-treatment tumour biopsies.

1. Signed written informed consent
2. ≥ 18 years old
3. All patients must have an activating KRAS mutation in tumour tissue samples from a prior test conducted by a clinical laboratory that has received international or country specific certification. Patients in Part B dosed on the basis of the local identification of an activating KRAS mutation, and whose KRAS mutation is not confirmed by the central laboratory (with the exception of locally obtained KRAS mutation status obtained from the approved tests), will remain on study but may be excluded from pharmacodynamic and anti-tumour activity analyses and replaced at the Sponsor's discretion. KRAS mutations identified in ctDNA (circulating tumour DNA) from blood are not acceptable; only mutations identified from tumour tissue are acceptable. Activating mutations may include but are not limited to:

   NSCLC KRAS mutations in codons G12/13, Q61, and A59

   mCRC KRAS mutations in codons G12/13 (Exon 2), Q61, A59 (Exon 3), K117, and A146 (Exon 4)

   Patient must agree to the collection of archival tumour tissue sample for biomarker analysis. If an archived tumour sample is not available a fresh tumour biopsy can be used.
4. Adequate organ system function as indicated by:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   2. Platelets ≥ 100 x 10^9/L
   3. Haemoglobin ≥ 9g/dL
   4. Activated partial thromboplastin time (aPTT) ≤ 1.5 times the upper limit of normal (ULN)
   5. Total bilirubin ≤ 1.5 mg/dL
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 times the ULN if no liver involvement or ≤ 5 times the ULN with liver involvement.
   7. Creatinine ≤ 1.5 times the ULN or creatinine clearance ≥ 60 mL/min as calculated by the Cockcroft-Gault method, or 24 hour measured urine creatinine clearance ≥ 60 mL/min.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Life expectancy ≥ 12 weeks
7. Male patients with female partners of child-bearing potential must be willing to use one highly effective form of contraception and must use a condom during their participation in this study and for 7 months following the last dose of the study drug. Male patients must refrain from donating sperm during their participation in the study and at least for 7 months after the last treatment.
8. Female patients must use a highly effective contraceptive measure from screening until 18 weeks after the last dose of drug. All methods of contraception (with the exception of total abstinence) should be used in combination with the use of a condom by a male sexual partner for intercourse. Female patients should not be breast-feeding and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

Post-menopausal women defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatment.

Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.

Exclusion Criteria:

1. Patients who have received chemotherapy, radiotherapy, hormonal therapy, immunotherapy or investigational drugs within 21 days or 5 half lives (whichever is shorter) from enrolment.
2. With the exception of alopecia, any unresolved toxicities from prior therapy greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of enrolment.
3. Unresolved immunotherapy-related hepatotoxicity from previous therapy.
4. Major surgery (excluding placement of vascular access) ≤ 21 days from beginning of the enrolment or minor surgical procedures ≤ 7 days. No waiting is required following implantable port and catheter placement.
5. Patients receiving full-dose anti-coagulation therapies.
6. Has active or prior documented autoimmune disease within the past 2 years with the exception of vitiligo, Grave's disease, and/or psoriasis not requiring systemic treatment.
7. Has a history of atypical Haemolytic Uremic Syndrome.
8. Patients with leptomeningeal metastases.
9. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 3 weeks prior to enrolment and there is no evidence of central nervous system disease progression or mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
10. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
11. Any of the following cardiac criteria:

    1. Congestive heart failure (CHF) per New York Heart Association (NYHA) classification > Class II.
    2. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
    3. Unstable angina or new-onset angina.
    4. QT interval (QTcF) >470 ms on screening electrocardiogram (ECG) by Fridericia's formula.
12. History of hypersensitivity to active or inactive excipients of AZD4785 or drugs with a similar chemical structure or class to AZD4785.
13. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
14. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Minimum of 28 days for a patient
  Determined through the evaluation of dose-limiting toxicity (DLT), adverse events, clinical laboratory test results, clinical evaluation and patient reported symptoms

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of AZD4785 | Samples for determination of AZD4785 plasma conc. will be collected at multiple times on Day 1 Cycle 1, pre-dose on Days 3, 5, and 8 of Cycle 1, Day 22 of Cycle 2, and Day 1 of Cycles 3 and 4. Time points may be adjusted based on emerging data.
  The concentration of AZD4785 in plasma, including peak concentration (Cmax), will be determined.
Area under the plasma concentration versus time curve (AUC) for AZD4785 | Samples for determination of AZD4785 plasma conc. will be collected at multiple times on Day 1 Cycle 1, pre-dose on Days 3, 5, and 8 of Cycle 1, Day 22 of Cycle 2, and Day 1 of Cycles 3 and 4. Time points may be adjusted based on emerging data.
  The concentration of AZD4785 in plasma, including area under the plasma concentration versus time curve (AUC), will be determined.
Objective Clinical Response | Every 8 weeks up to 12 months.
  CT scan to measure tumour
KRAS messenger RNA (mRNA) | 1-3 months
  Change from baseline in KRAS mRNA following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik-Tobias Arkenau, MD, Principal Investigator — Sarah Cannon Research Institute United Kingdom
Locations (5):
- United States (3):
  - Research Site, Sarasota, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Nashville, Tennessee
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search